CLINICAL TRIAL: NCT00818545
Title: Transcriptomic Study of ER 4017 Topical Application in Elderly Subject
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L'Oreal (Industry)
Responsible Party: Dr Tancrede and Pr L. Dubertret, Hôpital Saint-Louis, Centre de Recherche Bioclinique (CRB)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CRB-ER4017-07-01
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Aging
Keywords: aging; barrier function; transcriptomic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: ER4017 (hydroxypropyltetrahydropyrantriol); Drug: placebo
- hydroxypropyltetrahydropyrantriol (Experimental)
  Interventions: Drug: ER4017 (hydroxypropyltetrahydropyrantriol)

INTERVENTIONS:
Drug: ER4017 (hydroxypropyltetrahydropyrantriol) — Cream, 10%, each day during 3 months
  Other Names: ER4017
Drug: placebo
  Arms: 2

SUMMARY:
The stratum corneum (SC) is the superficial layer of the epidermis situated at the interface between the body and its outside environment. Its strategic position confers it a crucial role of protection against aggressions. After disruption, the kinetic of cutaneous barrier is slower in elderly comparatively to young subjects.

The purpose of this study is to investigate, by characterizing molecular events, the effectiveness of ER4017 (Hydroxypropyltetrahydropyrantriol) to restore kinetic barrier function after acute disruption of stratum corneum in ederly subjects.

10 male volunteers aged from 60 to 75 years are randomized to receive topical application of ER4017 versus placebo on skin inner forearms twice a day during 3 months. After sequential selloptape strips, epidermal samples of treated and control skin are removed under local anesthesia, using a dermatome. Differential gene expression analysis is performed using micro array techniques and quantitative RT-PCR.

treatment, randomized on the location, double blind, placebo control, internal control subject, prospective study.

DETAILED DESCRIPTION:
Structural modifications of the superficial dermis during the aging process associated to alterations in the GAG- and PG profile appear to impact the quality of the dermal epidermal junction (DEJ). Previous biological and clinical evaluations of ER4017, a C-glycoside biomimetic of xylose, showed its capacity to stimulate GAG- and PG synthesis and to improve morphogenesis of the whole DEJ.

The aim of the study is to investigate the gene expression in human epidermis treated with ER4017 following sequential sellotapes strips after a 3 months ER4017 topical application. For this purpose, the modulation of gene expression is determined using a cDNA microarray technology. Stratum corneum disruption is performed following 3 months topical application on skin inner forearms. All the experiments are performed in 10 elderly healthy men. Volunteers are clinically and biophysically evaluated at baseline and then at monthly intervals or at 3 months respectively.

ELIGIBILITY:
Inclusion Criteria:

* Phototype I to III
* Healthy skin on studied skin areas
* Subject having freely given his informed written consent.
* Cooperative subject, aware of the necessity to attend all the scheduled appointments during the study.
* Negative serology for HIV, hepatitis B and hepatitis C
* No past or present history of allergy linked either to one of the ingredients of the study cosmetic cream tested or to xylocaïne (anesthesia).

Exclusion Criteria:

* Cutaneous disease or previous malignant cutaneous lesion on the tested zones.
* Any treatment able to act on blood coagulation and homeostasis.

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Investigate the effectiveness of an anti aging topical treatment by characterizing molecular modifications linked to barrier function recovery following a disruption of stratum corneum. | day 0(visit selection), day 1 (inclusion visit), day 2 to day 84 (treatment period), day 85 (end of the treatment), day 92 and day 99 (follow up period)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Dubertret, Prof, Principal Investigator — centre de recherche bioclinique -Hopital st louis
Locations (1):
- Centre de recherche bioclinique -Hopital st louis, Paris, France